CLINICAL TRIAL: NCT07075276
Title: Injection of Liquid Phase Concentrated Growth Factor Versus Conventional Arthrocentesis in Management of Temporomandibular Disc Displacement: A Randomized Controlled Clinical Trial
Brief Title: Liquid Phase Concentrated Growth Factor Versus Conventional Arthrocentesis in Temporomandibular Disc Displacement
Acronym: LPCGF in TMDs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Horus University (Other)
Responsible Party: Principal Investigator, Mohamed Ali Habib, Teaching assistant, Horus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CGF for management of TMDs
Record Dates: First submitted 2025-07-11; First posted 2025-07-20 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Temporomandibular Disorders (TMD); Internal Derangement of the Tempromandibular Joint; Anterior Disc Displacement
Keywords: Temporomandibular disorder; Concentrated growth factor; Anterior disc displacement with reduction; Anterior disc displacement without reduction; Arthrocentesis
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Intervention Model Description: 16 patients with anterior disc displacement with or without reduction will be treated with liquid phase concentrated growth factor and 16 patients will be treated with conventional arthrocentesis
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 16 patients have anterior disc displacement with or without reduction will be treated with injection of liquid phase concentrated growth factor
  Interventions: Procedure: Liquid Phase Concentrated Growth Factor
- Group B (Active Comparator): 16 patients have anterior disc displacement with or without reduction will be treated with conventional arthrocentesis
  Interventions: Procedure: Conventional arthrocentesis

INTERVENTIONS:
Procedure: Liquid Phase Concentrated Growth Factor — 16 patients with anterior disc displacement with or without reduction randomly allocated to be treated with injection of liquid phase concentrated growth factor
  Arms: Group A
Procedure: Conventional arthrocentesis — 16 patients with anterior disc displacement with or without reduction randomly allocated to be treated with conventional arthrocentesis
  Arms: Group B

SUMMARY:
This study aims to rigorously assess the effectiveness of LPCGF in the management of internal disc displacement in patients with TMD through a randomized clinical trial. By comparing LPCGF therapy with conventional arthrocentesis, this research looks to provide robust evidence on the efficacy, safety, and potential role of (LPCGF) as an alternative therapeutic choice for IDD.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults aged 18-45 years. 2. Patients scored as (ASA I).9 3. Presence of complete or nearly complete set of natural dentition with Angle class I occlusion. 4. Diagnosed with unilateral involvement of disc displacement, according to the Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD).10 5. Symptoms include one or more of the following: pain, joint sounds, and limited mandibular movement (Maximum Mouth Opening< 40mm) 6. No prior surgical intervention for TMD. 7. Patient's willingness to participate and follow the study protocol.

Exclusion Criteria:

* 1. TMJ pathology related to mechanical deformities 2. Psychiatric problems or presence of systemic diseases that may affect healing (e.g., uncontrolled diabetes, autoimmune disorders, hematologic or neurologic disorders, inflammatory or connective tissue disorders as well as rheumatological or previous infectious diseases, head and neck cancer). 3. Patient unwilling or has contraindication to MRI 4. Previous injections or surgical interventions of the TMJ. 5. Concurrent use of anticoagulants or anti-inflammatory medications within the last 30 days. 6. Pregnant or breastfeeding women. 7. History of trauma or infection in the TMJ region. 8. Allergy to local anesthetics or other components used in the study. 9. Patients diagnosed with (Disc Displacement with reduction with no pain or limited mandibular movements).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Assess and comparing the pain of both groups | Assessed at baseline (before treatment),1week, 1 month, 3 months, and 6 months after the intervention.
  measured using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst pain)
Assess and comparing the mouth opening of both groups | Assessed at baseline (before treatment),1week, 1 month, 3 months, and 6 months after the intervention.
  measured in millimeters (Maximum inter-incisal opening measured by the distance in millimeters between the incisal edges of the upper and lower central incisors in vertical direction at maximum pain free mouth opening) by using caliper. and comparing the results of both groups

SECONDARY OUTCOMES:
Joint sounds | Assessed at baseline (before treatment),1week, 1 month, 3 months, and 6 months after the intervention.
  (clicking and crepitus) evaluated by clinical examination; presence of joint noise at opening and closing was evaluated by light bilateral digital palpation during jaw movement.
Mandibular deviation during mouth opening. | Assessed at baseline (before treatment),1week, 1 month, 3 months, and 6 months after the intervention.
  By clinical examination , observe mandibular deviation toward right or left side or deflection during opening and closing the mouth
Lateral and protrusive movements | Assessed at baseline (before treatment),1week, 1 month, 3 months, and 6 months after the intervention
  (Range of lateral and protrusive movements measured by the distance in millimeters between the upper and lower midlines in horizontal direction on lateral and protrusive movements by using caliper).
tenderness on palpation | Assessed at baseline (before treatment),1week, 1 month, 3 months, and 6 months after the intervention.
  Presence or absence of joint tenderness on palpation: recorded as tender or not tender.
TMD symptoms | Assessed at baseline (before treatment),1week, 1 month, 3 months, and 6 months after the intervention.
  TMD symptoms were evaluated using Modified Helkimo Index

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ali Habib, Teaching Assistant, Principal Investigator — Horus University in Egypt - Faculty of dentistry; Eman AbdElsalam Yousef, Ass. prof, Study Director — Horus University in Egypt- Faculty of dentistry; Ahmed Khalil, lecturer, Study Director — Horus University in Egypt - Faculty of dentistry
Locations (1):
- Faculty of Dentistry- Horus University in Egypt, Damietta, New Damietta, Egypt

IPD SHARING:
Plan to Share IPD: No